CLINICAL TRIAL: NCT01121237
Title: An International, Prospective, Open-label, Multicenter, Pharmacoepidemiological Study to Determine Predictors of Clinical Outcomes in Haemodialysis Patients With Anaemia Treated With Biosimilar Epoetin Alfa
Brief Title: MONITOR-CKD5 - Multi-level Evaluation of Anaemia Treatment, Outcomes, and Determinants in Chronic Kidney Disease Stage 5
Acronym: MONITOR-CKD5
Status: Completed | Type: Observational
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HX575-503
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Kidney Disease; End-stage Renal Disease; Anaemia
Keywords: chronic kidney disease; end-stage renal disease; renal anaemia; epoetin alfa
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Anemia | interventions — Biosimilar Pharmaceuticals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CKD5, renal anaemia, haemodialysis: CKD5, renal anaemia, haemodialysis receiving recombinant human erythropoietin alfa (biosimilar)
  Interventions: Drug: Recombinant human erythropoietin alfa (biosimilar)

INTERVENTIONS:
Drug: Recombinant human erythropoietin alfa (biosimilar) — Recombinant human erythropoietin alfa (biosimilar) commercially available as prescribed per treating physician
  Other Names: biosimilar epoetin alfa

SUMMARY:
MONITOR-CKD5 is an observational, pharmaco-epidemiological study to evaluate the multi-level factors and outcomes associated with the treatment of renal anaemia with biosimilar epoetin alfa in Stage 5 CKD patients requiring haemodialysis.

DETAILED DESCRIPTION:
See the following publication:

Gesualdo, L., London, G., Turner, M., Lee, C., MacDonald, K., Covic, A., Zaoui, P., Combe, C., Dellana, F., Muenzberg, M., & Abraham, I. (in press). A pharmacoepidemiological study of the multi-level determinants, predictors, and clinical outcomes of biosimilar epoetin alfa for renal anemia in hemodialysis patients: background and methodology of the MONITOR-CKD5 study. Internal and Emergency Medicine. (DOI 10.1007/511739-011-0622-7)

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (age > 18 years).
* On chronic haemodialysis due to end-stage renal disease (CKD5) of original or grafted kidneys for any duration.
* Diagnosed with renal anaemia; i.e., anaemia due to impaired production of endogenous erythropoietin secondary to kidney failure.
* Treated with commercially available intravenous EPOETIN ALFA HEXAL® per physician's best clinical judgment and under consideration of available guidance and evidence.
* Female patients must be either post-menopausal for one year or surgically sterile or using effective contraceptive methods such as barrier method with spermicide or an intra-uterine device. Oral contraceptive use is allowed.
* Informed written consent to participate in the study by patients or their legal guardian.

Exclusion Criteria:

* Known sensitivity to EPOETIN ALFA HEXAL® or any other ESA.
* Solid or hematological neoplasia being treated with chemotherapy.
* Treatment with any myelosuppressant medications.
* Blood transfusion dependency.
* History of pure red cell aplasia.
* Bleeding episode in 30 days prior to enrollment.
* Orthopaedic surgery in 30 days prior to enrollment.
* Patients with several medical condition(s) that in view of the investigator prohibits participation in the study.
* Patients with willfully negligent nonadherence to their haemodialysis, medication, nutrition, and/or other recommended treatment regimens.
* Use of any investigational agent in the 30 days prior to enrollment.
* Women of childbearing potential not using the contraception method(s) described above.
* Women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease stage 5 with renal anemia and on haemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 2086 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Haemoglobin outcomes, including haemoglobin levels in g/dL, change in haemoglobin levels over time (in g/dL and %), number and proportion of patients with haematopoietic response, number and proportion of patients reaching target haemoglobin levels. | every month for 24 months

SECONDARY OUTCOMES:
Number and proportion of participants with thrombovascular events, hospitalization,and mortality as measures of safety. | Every month for 24 months + as occurring between visits
  Safety will be assessed every month for 24 months. In addition, any safety events reported by the patient or observed by clinicians in-between the monthly assessments will be recorded at the time of report or occurrence, and will be addressed at that time as necessary.

CONTACTS AND LOCATIONS:
Overall Officials: HEXAL AG, Study Chair — Hexal AG
Locations (95):
- Austria (5):
  - Sandoz Investigational Site, Bregenz
  - Sandoz Investigational Site, Eisenstadt
  - Sandoz Investigational Site, Feldkirch
  - Sandoz Investigational Site, Nenzing
  - Sandoz Investigational Site, Vienna
- France (5):
  - Sandoz Investigational Site, Ajaccio
  - Sandoz Investigational Site, Dourlers
  - Sandoz Investigational Site, Fourmies
  - Sandoz Investigational Site, Lille
  - Sandoz Investigational Site, Saint-Quentin
- Germany (37):
  - Sandoz Investigational Site, Alsfeld
  - Sandoz Investigational Site, Arnstadt
  - Sandoz Investigational Site, Bad Neustadt A. D. Saale
  - Sandoz Investigational Site, Bassum
  - Sandoz Investigational Site, Berlin
  - Sandoz Investigational Site, Bochum
  - Sandoz Investigational Site, Cloppenburg
  - Sandoz Investigational Site, Cochem
  - Sandoz Investigational Site, Darmstadt
  - Sandoz Investigational Site, Dresden
  - Sandoz Investigational Site, Duisburg
  - Sandoz Investigational Site, Düsseldorf
  - Sandoz Investigational Site, Erftstadt
  - Sandoz Investigational Site, Georgsmarienhütte
  - Sandoz Investigational Site, Greifswald
  - Sandoz Investigational Site, Güstrow
  - Sandoz Investigational Site, Herne
  - Sandoz Investigational Site, Herzberg
  - Sandoz Investigational Site, Hoyerswerda
  - Sandoz Investigational Site, Höchstadt an der Aisch
  - Sandoz Investigational Site, Kamen
  - Sandoz Investigational Site, Kiel
  - Sandoz Investigational Site, Magdeburg
  - Sandoz Investigational Site, Mettmann
  - Sandoz Investigational Site, Munich
  - Sandoz Investigational Site, Nuremberg
  - Sandoz Investigational Site, Osnabrück
  - Sandoz Investigational Site, Pinneberg
  - Sandoz Investigational Site, Quedlinburg
  - Sandoz Investigational Site, Remagen
  - Sandoz Investigational Site, Rendsburg
  - Sandoz Investigational Site, Schrobenhausen
  - Sandoz Investigational Site, Schwabach
  - Sandoz Investigational Site, Seehausen
  - Sandoz Investigational Site, Viersen
  - Sandoz Investigational Site, Wetzlar
  - Sandoz Investigational Site, Wilhelmshaven
- Italy (18):
  - Sandoz Investigational Site, Acireale
  - Sandoz Investigational Site, Altamura
  - Sandoz Investigational Site, Arenzano
  - Sandoz Investigational Site, Arezzo
  - Sandoz Investigational Site, Biella
  - Sandoz Investigational Site, Catania
  - Sandoz Investigational Site, Chivasso
  - Sandoz Investigational Site, Cinisello Balsamo
  - Sandoz Investigational Site, Cirié
  - Sandoz Investigational Site, Cosenza
  - Sandoz Investigational Site, Cuneo
  - Sandoz Investigational Site, Ivrea
  - Sandoz Investigational Site, Montevarchi
  - Sandoz Investigational Site, Pavia
  - Sandoz Investigational Site, Pontecorvo
  - Sandoz Investigational Site, Putignano
  - Sandoz Investigational Site, Roma
  - Sandoz Investigational Site, Torino
- Poland (7):
  - Sandoz Investigational Site, Bialystok
  - Sandoz Investigational Site, Ciechanów
  - Sandoz Investigational Site, Gdansk
  - Sandoz Investigational Site, Lublin
  - Sandoz Investigational Site, Poznan
  - Sandoz Investigational Site, Rzeszów
  - Sandoz Investigational Site, Wołomin
- Romania (9):
  - Sandoz Investigational Site, Bistriţa
  - Sandoz Investigational Site, Brasov
  - Sandoz Investigational Site, Brăila
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Miercurea-Ciuc
  - Sandoz Investigational Site, Odorheiu Secuiesc
  - Sandoz Investigational Site, Reşiţa
  - Sandoz Investigational Site, Roman
  - Sandoz Investigational Site, TG. Jiu
- Slovenia (2):
  - Sandoz Investigational Site, Maribor
  - Sandoz Investigational Site, Šempeter pri Gorici
- Spain (4):
  - Sandoz Investigational Site, Ávila
  - Sandoz Investigational Site, León
  - Sandoz Investigational Site, Seville
  - Sandoz Investigational Site, Zamora
- Switzerland (4):
  - Sandoz Investigational Site, Fribourg
  - Sandoz Investigational Site, Lausanne
  - Sandoz Investigational Site, Nyon
  - Sandoz Investigational Site, Zurich
- United Kingdom (4):
  - Sandoz Investigational Site, Cambridge
  - Sandoz Investigational Site, Chester
  - Sandoz Investigational Site, Norwich
  - Sandoz Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Combe C, Mann J, Goldsmith D, Dellanna F, Zaoui P, London G, Denhaerynck K, Krendyukov A, Abraham I, MacDonald K. Potential life-years gained over a 5-year period by correcting DOPPS-identified modifiable practices in haemodialysis: results from the European MONITOR-CKD5 study. BMC Nephrol. 2019 Mar 5;20(1):81. doi: 10.1186/s12882-019-1251-z. PMID 30836953
- [Derived] Gesualdo L, London G, Turner M, Lee C, Macdonald K, Goldsmith D, Covic A, Zaoui P, Combe C, Mann J, Dellanna F, Muenzberg M, Abraham I. A pharmacoepidemiological study of the multi-level determinants, predictors, and clinical outcomes of biosimilar epoetin alfa for renal anaemia in haemodialysis patients: background and methodology of the MONITOR-CKD5 study. Intern Emerg Med. 2013 Aug;8(5):389-99. doi: 10.1007/s11739-011-0622-7. Epub 2011 May 18. PMID 21590439